CLINICAL TRIAL: NCT06575387
Title: The Utility of Partogram in Management of Active Labor in Primigravidae and Its Impact In Qena Governorate
Brief Title: The Utility of Partogram in Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Collaborators: Al-Azhar University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Manal Ahmed Mohamed
Record Dates: First submitted 2024-08-25; First posted 2024-08-28 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2023-09

CONDITIONS: Labor Onset

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Uncomplicated Normal Labour (Active Comparator): About 140 prime gravidae females delivered before or at alert line
  Interventions: Procedure: Partogram
- Group B: Complicated Normal Labour (Active Comparator): About 40 prime gravidae females delivered between alert and action line
  Interventions: Procedure: Partogram
- Group C: Cesarean Section Labour (Active Comparator): About 20 prime gravidae females delivered after action line
  Interventions: Procedure: Partogram

INTERVENTIONS:
Procedure: Partogram — to evaluate the utility of partogram in management and progress of active labor in Primigravidae.

SUMMARY:
The partograph serves as "early warning system" and it has shown to be effective in preventing prolonged labour, in reducing operative interventions and in improving the neonatal outcome.

"A picture is worth a thousand words". A partograph review if well recorded provides rapid and comprehensive information about progress of labour when compared with a review of detailed handwritten case sheets. Partograph is a Latin/Greek hybrid word synonymous with parturition recorded in a graphic form.

DETAILED DESCRIPTION:
labour is a natural physiological process characterized by progressive increase in the frequency, intensity and duration of uterine contractions, resulting in effacement and dilatation of the cervix with descent of the foetus through the birth canal. This physiological process may take time lead to pathological one and failure to recognize this would result in prolonged labour with the resultant increase in the intensity in the morbidity and mortality of both foetus and the mother.This leads to surgical intervention with further danger to both the mother and foetus. Hence, prolonged labour and obstructed labour must be prevented by timely and effective measures, so as to give the mother a safe and happy experience of labour and child birth. The safe mother hood initiative (SMI) emphasises that the monitoring of labour for early detection of dystocia is one of the most important approaches for reducing maternal and neonatal morbidity and mortality.

In this context, the partogram has been adopted by the WHO (World health Organization) to monitor labour in maternity clinics in developing countries as a simple managerial tool to prevent prolonged labour, obstructed labour and its sequelle. The paperless partograph refers to monitoring progress of labour and reaching to an accurate decision for intervention to ensure safe delivery.

The partograph, a graphic recording of progress of labour and salient features in the mother and foetus has been used to detect labour that is not progressing normally, to help in early decision on augmentation and termination of labour.

WHO partograph is a composite graphic representation of events that takes place in labour plotted against time in hours on a pre-printed paper. It consists of three parameters:

ELIGIBILITY:
Inclusion Criteria:

* Primigravida, 20 and 35 years old
* Gestational age 37 - 41 weeks with vertex presentation
* Singleton pregnancy
* Spontaneous or induced labour
* First stage of labour with cervical dilatation < than 7 cm.

Exclusion Criteria:

* Abnormal presentation
* Macrosomic baby
* Contacted pelvis
* Multifetal gestations
* Antepartum haemorrhage
* Cases with high risk pregnancy as Severe PIH, Severe anaemia and gestational diabetes mellitus.
* Patient refused to enrolled in the research

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Mode of Delivery | 24 hours
  The mode of delivery was assessed by the condition of the mother and the fetus by BISHOP score (The Bishop score is a cervical assessment system used to predict the success of labor induction. This scoring system evaluates several clinical parameters of the cervix, including dilation, effacement, position, consistency, and the fetal head's station in the pelvis).

CONTACTS AND LOCATIONS:
Overall Officials: Abd El-Aziz Galal El-Din El-Darwish, Professor, Study Chair — Al-Azhar University, Faculty of medicine, Assuit.; Khaled Mohamed Ahmed M. Abdallah, Assist.Professor, Study Director — Al-Azhar University, Faculty of medicine, Assuit.
Locations (1):
- Al-Azhar University hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided